CLINICAL TRIAL: NCT00187512
Title: SCOPE: Observational Study of the Consequences of the Protease Inhibitor Era
Acronym: SCOPE
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-01330
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections
Keywords: HIV; Antiretroviral Agents; Drug Resistance, Multiple; Long Term Non Progression; Long Term Non Progressor; Elite Suppression; Elite Suppressor; Natural History; Observational
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, PMBCs, saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
SCOPE is an observational, prospective study of HIV-1 infected volunteers designed to provide a specimen bank of samples with carefully characterized clinical data. SCOPE specimens will be used to examine multiple questions involving virologic, immunologic, and host factors involved in HIV-1 infection, progression, non-progression, response to treatment, control of HIV-1 virus, and evolution of drug resistance.

DETAILED DESCRIPTION:
SCOPE is an observational, prospective study of HIV-1 infected volunteers designed to provide a specimen bank of samples with carefully characterized clinical data. Samples from SCOPE will be used to examine:

1. Virologic, immunologic, and host factors involved in the natural control of HIV-1 infection (long term non-progression and/or virologic control of HIV-1 without antiretroviral therapy)
2. Virologic and immune correlates associated with disease progression
3. Evolution of antiretroviral drug resistance
4. Factors associated with transmission or acquisition of HIV infection

Enrolled subjects are seen at San Francisco General Hospital every four months for a detailed interview, saliva collection, and blood draw. Baseline visits take approximately one hour, follow up visits take approximately 20-40 minutes. No personal identifiers are used for specimen bank samples.

ELIGIBILITY:
Inclusion Criteria:

SCOPE is currently recruiting HIV-1 infected subjects with any of the following criteria:

1. Documented HIV viral load less than 2000 copies/ml WITHOUT taking antiretroviral therapy
2. Undetectable HIV viral load with CD4 T-cells consistently less than 350 for the last 12 months while taking a stable antiretroviral regimen.
3. Antiretroviral naive and planning to start an antiretroviral regimen - any CD4 or HIV viral load acceptable.
4. Long-term Non Progressors: HIV-positive at least 10 years, no antiretroviral therapy for the past 10 years or more, any viral load acceptable, CD4-T cell count always above 500.

Exclusion Criteria:

1. Active opportunistic infection or systemic treatment for opportunistic infection within the last 4 months (oral candidiasis acceptable)
2. Active treatment for cancer
3. Active treatment for hepatitis C requiring interferon based therapy
4. Immunosuppressive therapy taken within the last 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is open to eligible subjects who are able to perform study visits at San Francisco General Hospital or the San Francisco VA Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2000-03; Primary Completion 2032-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
The general theme of this core is to investigate the relationship between the virologic response to antiretroviral therapy and clinical outcome. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Steven G. Deeks, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Favre D, Stoddart CA, Emu B, Hoh R, Martin JN, Hecht FM, Deeks SG, McCune JM. HIV disease progression correlates with the generation of dysfunctional naive CD8(low) T cells. Blood. 2011 Feb 17;117(7):2189-99. doi: 10.1182/blood-2010-06-288035. Epub 2011 Jan 3. PMID 21200021